CLINICAL TRIAL: NCT05050526
Title: Effects of a Real-time Videoconference-based Exercise Program in Eldercare Workers: a Randomized Controlled Trial
Brief Title: Real-time Videoconference-based Exercise in Eldercare Workers
Acronym: ReViEEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ander Espin (Other)
Collaborators: Caser Residencial Betharram (Unknown); Fundación Aspaldiko (Unknown); Grupo Servicios Sociales Integrados (Unknown); Igurco Residencias Sociosanitarias (Unknown); Grupo Colisée (Unknown)
Responsible Party: Sponsor-Investigator, Ander Espin, Predoctoral Researcher, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Eldercare2021
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pain; Mental Disorders
Keywords: Eldercare; Caregiver; Exercise; Tele-health; Musculoskeletal disorders; Mental disorders; Absenteeism; Work ability; Work performance
MeSH Terms: conditions — Pain; Mental Disorders; Motor Activity; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators in charge of doing the statistical analysis and assessing the outcome measures (e.g., physical performance tests) will be blinded to group allocation. Due to the characteristics of the study, blinding of the participants (i.e., eldercare workers) and the care provider (i.e., professional conducting the exercise sessions) to the group allocation is not possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise program (Experimental): Participants in the experimental group will take part in a 12-week exercise program.
  Interventions: Behavioral: Real-time videoconference-based Exercise program
- Control (No Intervention): Participants in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Real-time videoconference-based Exercise program — 12-week exercise program consisting of two weekly 45 minute group-based sessions, remotely supervised by a professional via real-time videoconference. Each session will consist of a warm-up (5-10 min), general strengthening (30 min) and cool-down (5-10 min). Warm-up will include general joint mobility and exercises focused on increasing heart rate. General strengthening will include 4 series of 6 exercises (2 for lower limb, 2 for upper limb and 2 for the trunk) performed with minimal equipment, combining body-weight and elastic-band exercises. Three difficulty levels will be set for each of the exercises, and progression will be made at weeks 5 and 9. Participants will be asked to work in a given rate of perceived exertion (between 3 and 5 in Borg's CR10 scale) and not to reach failure in any of the exercises. Cool-down will include stretching and breathing/relaxing exercises.
  Arms: Exercise program

SUMMARY:
Formal caregiving of elderly dependent people is a both physically and psychologically demanding job, and both musculoskeletal and mental disorders with a negative impact in general health and quality of life are habitual among eldercare workers. Previous research has shown that physical exercise programs can reduce and/or prevent those disorders, consequently improving well-being at work.

Online exercise interventions might be a cost-effective tool, as they can reach a large number of people at a relatively low cost. Moreover, they are compatible with situations in which interpersonal physical distancing is required, such as the current COVID-19 pandemic. However, real-time videoconference-based exercise interventions have not yet been studied in working populations.

Thus, the aim of this study is to assess the effects of a real-time videoconference-based exercise intervention in eldercare workers. The primary outcome will be low back pain. Pain in neck, shoulders and wrists/hands will also be recorded, as well as additional measures of physical fitness, psychoaffective state, health and work-related variables. All outcomes will be measured at baseline and at 12-week and 48-week follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Professional eldercare workers with ≥3 months of experience in the profession
* Employment contract at least until the anticipated date of study end

Exclusion Criteria:

* Pregnancy
* Contraindication to exercise according to the American College of Sports Medicine Guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline average pain intensity at 12 weeks | At baseline and at 12-week follow-up
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline average pain intensity at 48 weeks | At baseline and at 48-week follow-up
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline highest pain intensity at 12 weeks | At baseline and at 12-week follow-up
  Highest pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline highest pain intensity at 48 weeks | At baseline and at 48-week follow-up
  Highest pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline pain frequency at 12 weeks | At baseline and at 12-week follow-up
  Number of days in pain during the last 7 days (0-7). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline pain frequency at 48 weeks | At baseline and at 48-week follow-up
  Number of days in pain during the last 7 days (0-7). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline pain interference at 12 weeks | At baseline and at 12-week follow-up
  Number of days in which pain negatively interferes with work during the last 7 days of work (0-7). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.
Change from baseline pain interference at 48 weeks | At baseline and at 48-week follow-up
  Number of days in which pain negatively interferes with work during the last 7 days of work (0-7). This information will be collected for pain in the low back, neck, shoulders and wrists/hands.

SECONDARY OUTCOMES:
Analgesic medication consumption frequency | At baseline and at 12-week and 48-week follow-ups
  Number of days in which analgesic medication is taken during the last 7 days (0-7).
5-repetition sit-to-stand test | At baseline and at 12-week and 48-week follow-ups
  It measures lower limb strength based on the time taken by the participant to get up from and sit down on a chair five times as quickly as possible.
Kneeling push-up test | At baseline and at 12-week and 48-week follow-ups
  It measures upper limb strength based on the maximum number of "knee push-ups" the participant can perform until failure.
Shirado-Ito trunk flexor endurance test | At baseline and at 12-week and 48-week follow-ups
  It measures trunk flexor endurance based on the maximum time the participant is able to maintain a defined body position, which mainly activates trunk flexor muscles.
Subjective Happiness scale | At baseline and at 12-week and 48-week follow-ups
  It is comprised of 4 items, each of them answered with a score between 1 and 7. A single composite score is obtained by averaging the responses to the 4 items, and a higher score corresponds to a greater happiness.
Goldberg Anxiety and Depression scale | At baseline and at 12-week and 48-week follow-ups
  The scale includes 9 items for anxiety symptoms and 9 items for depression symptoms. Each item is answered with a "Yes" or a "No". A higher number of positive answers corresponds to a higher risk of suffering a clinically relevant anxiety or depression disorder, respectively.
Maslach Burnout Inventory | At baseline and at 12-week and 48-week follow-ups
  The Inventory is comprised of 22 items corresponding to three domains: personal accomplishment, emotional exhaustion and depersonalization. Each item is answered in a 0-6 Likert scale depending on the frequency with which the participant experiences the feelings described. One total score per domain is obtained.
Single-Item Sleep Quality Scale | At baseline and at 12-week and 48-week follow-ups
  It evaluates overall sleep quality in the last 7 days with a numerical scale that ranges between 0 (terrible) and 10 (excellent).
Hypnotic/anxiolytic medication consumption frequency | At baseline and at 12-week and 48-week follow-ups
  Number of days in which hypnotic/anxiolytic medication is taken during the last 7 days (0-7).
EuroQol-5D 0-100 health state scale | At baseline and at 12-week and 48-week follow-ups
  It measures self-perceived current health state in a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Work Ability | At baseline and at 12-week and 48-week follow-ups
  Work ability will be assessed by the following item extracted from the Workability Index: "assuming that your work ability at its best has a value of 10 points, how many points would you rate your current work ability?". Participants are asked to give a score ranging from 0 (completely unable to work) to 10 (lifetime best work ability).
Work Performance | At baseline and at 12-week and 48-week follow-ups
  Work performance will be assessed by the following item extracted from the World Health Organization Health and Work Performance Questionnaire: "On a scale from 0 to 10 where 0 is the worst job performance anyone could have at your job and 10 is the performance of a top worker, how would you rate your overall work performance on the days you worked during the last 12 weeks?" Participants are asked to give a score between 0 and 10.
Borg's CR-10 scale for perceived physical exertion at work | At baseline and at 12-week and 48-week follow-ups
  It measures perceived physical exertion while doing physical work in a scale ranging from 0 (nothing at all) to 10 (extremely strong).
Absenteeism | At baseline and at 12-week and 48-week follow-ups
  Days of absence from work during the last year will be collected from the official registry of the company and by self-reported questionnaire. Presence of absenteeism (yes/no), days of absence (n) and reason will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Ander Espin, PhD Student, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (2):
- Spain (2):
  - Residencia Aspaldiko, Portugalete, Bizkaia
  - Caser Residencial Betharram, Hondarribia, Gipuzkoa

REFERENCES:
- [Background] Espin A, Irazusta J, Segovia Celaya I, Mosquera Lajas A, Gonzalez-Templado V, Rodriguez-Larrad A. Effects of a videoconference-based therapeutic exercise intervention on the musculoskeletal pain of eldercare workers: protocol for the ReViEEW randomized controlled trial. BMC Musculoskelet Disord. 2023 Jun 6;24(1):463. doi: 10.1186/s12891-023-06584-7. PMID 37280584
- [Result] Espin A, Irazusta J, Aiestaran M, Latorre Erezuma U, Garcia-Garcia J, Arrinda I, Acedo K, Rodriguez-Larrad A. Videoconference-Supervised Group Exercise Reduces Low Back Pain in Eldercare Workers: Results from the ReViEEW Randomised Controlled Trial. J Occup Rehabil. 2025 Mar;35(1):66-77. doi: 10.1007/s10926-024-10182-2. Epub 2024 Apr 17. PMID 38632115
- [Derived] Espin A, Rodriguez-Larrad A, Ruiz-Fernandez A, Martin-Perez A, Fernandez-Gutierrez N, Andersen LL, Irazusta J. Predictors of response to physical exercise for low back pain: a secondary analysis of the ReViEEW trial. Musculoskelet Sci Pract. 2026 Feb;81:103465. doi: 10.1016/j.msksp.2025.103465. Epub 2025 Dec 3. PMID 41353795
- [Derived] Espin A, Irazusta J, Urquiza M, Ruiz-Fernandez A, Latorre Erezuma U, Collado Torres L, Andersen LL, Rodriguez-Larrad A. Videoconference-Supervised Exercise for Low Back Pain in Eldercare Workers: One-Year Follow-up of the ReViEEW Randomized Controlled Trial. J Occup Environ Med. 2025 Oct 1;67(10):e720-e728. doi: 10.1097/JOM.0000000000003474. Epub 2025 Jun 2. PMID 40561221
- See also: Link to study protocol published in BMC Musculoskeletal Disorders — https://pubmed.ncbi.nlm.nih.gov/37280584/
- See also: Link to study 12-week results in the Journal of Occupational Rehabilitation — https://pubmed.ncbi.nlm.nih.gov/38632115/